CLINICAL TRIAL: NCT06925373
Title: Housing, Environment, And Living Conditions for Transformed Health (HEALTHe Birmingham)
Brief Title: Housing, Environment, And Living Conditions for Transformed Health
Acronym: HEALTHe
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Gabriela R Oates, Associate Professor, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB-300013400; 1U01NR021591 (NIH)
Record Dates: First submitted 2025-03-11; First posted 2025-04-13 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Lung Diseases; Chronic Disease
Keywords: Lung Health; Chronic Disease
MeSH Terms: conditions — Lung Diseases; Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Elyton Village Community (Active Comparator): Participants will receive improved neighborhood environment (built and social) and indoor air purification.
  Interventions: Other: Indoor Air Purification; Other: Neighborhood Improvements
- Southtown Court Community (Active Comparator): Participants will receive new public housing.
  Interventions: Other: Housing Improvements
- Smithfield Court Community (Active Comparator): Participants will receive new public housing and improved neighborhood environment (built and social).
  Interventions: Other: Neighborhood Improvements; Other: Housing Improvements
- Collegeville Community (Active Comparator): Participants will receive indoor air purification.
  Interventions: Other: Indoor Air Purification

INTERVENTIONS:
Other: Indoor Air Purification — An indoor air purifier with a dual HEPA/activated carbon filter, a usage tracker, and an indoor air quality monitor will be installed in public housing residences.
  Other Names: Coway Airmega 400
  Arms: Collegeville Community; Elyton Village Community
Other: Neighborhood Improvements — Improved built environment (green space, sidewalks, street lights) and social environment (educational and workforce development programs, wrap-around social services, Internet access).
  Arms: Elyton Village Community; Smithfield Court Community
Other: Housing Improvements — High-quality public housing
  Arms: Smithfield Court Community; Southtown Court Community

SUMMARY:
This project will compare the health effects of public housing renovation, neighborhood built and social environment improvements, and indoor air purification, alone and in combination, as well as the cost effectiveness of each approach.

STUDY 1: The study will assess the effects of public housing and neighborhood environment (built and social) improvements on health-related behaviors, psychosocial and physiologic stress, and self-reported and physiological markers of lung health and chronic disease.

STUDY 2: The study will determine whether indoor air purification can positively impact lung health in public housing sites not undergoing housing renovation, comparing a site near industrial pollution vs one less contaminated.

DETAILED DESCRIPTION:
Participants will complete surveys, physical exam, lung function tests, and blood draw. An indoor air purifier with a usage tracker and an indoor air quality monitor will be provided, and used filters will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 years and older
* English speaking
* Residents of one of 4 public housing site in Birmingham, Alabama

Exclusion Criteria:

* Individuals who are not 18 years or older
* Do not speak English
* Do not meet the residency criteria

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2025-06-18 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Change in Patient-Reported Outcomes Measurement Information System (PROMIS-10) Global Health | Baseline, 12 months, 24 months
  A self-reported measure of physical, mental, and social health. 10 item questionnaire T-score metric from zero to 100 where higher T-scores indicate better health.
Change in Allostatic load | Baseline, 12 months
  Measure of cumulative stress burden as the number of 10 indicators above a threshold: (1) serum albumin <3.8 g/dL, (2) C Reactive Protein (CRP) >3 mg/L, (3) High-Density Lipoprotein (HDL) <40 mg/dL, (4) total cholesterol ≥240 mg/dL, (5) heart rate ≥90 beats/min, (6) systolic Blood Pressure (BP) ≥140 mmHg, (7) diastolic BP ≥90 mmHg, (8) serum creatinine ≥1.3 mg/dL, (9) Blood Urea Nitrogen (BUN) ≥18 mg/dL, and (10) waist circumference >88 cm in women, >102 cm in men.
Change in Indoor Air Quality | Baseline, 6 months, 12 months (Study 2 only)
  Particulate matter (PM2.5). Measures particles in the air that are 2.5 micrometers or smaller in diameter.

SECONDARY OUTCOMES:
The percentage change in FEV1/FVC | Baseline, 6 months, 12 months (Study 2 only)
  FEV1/FVC. A measure of lung funtion that compares the amount of air exhaled in the first second (FEV1) to the total amount of air exhaled in a forced breath (FVC).

CONTACTS AND LOCATIONS:
Overall Officials: Gabriela R Oates, PhD, Principal Investigator — University of Alabama at Birmingham (UAB)
Locations (1):
- UAB Lung Health Center, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the reported results, after de-identification.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available beginning 12 months and ending 36 months after publication.
Access Criteria: Data will be available to investigators who submit an approved proposal and sign a Data Use Agreement. Proposals should be submitted to goates@uab.edu.